CLINICAL TRIAL: NCT06848491
Title: Using Tailored mHealth Strategies to Promote Weight Management Among Adolescent and Young Adult Cancer Survivors (AYA Well)
Brief Title: Using Tailored mHealth Strategies to Promote Weight Management Among Adolescent and Young Adult Cancer Survivors
Acronym: AYAWell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Virginia Commonwealth University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCCC2318; 5R01CA270111 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Cancer; Physical Activity; Cancer Survivorship; Diet
MeSH Terms: conditions — Obesity; Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions following baseline assessments in a 1:1 ratio. The conditions are Intervention or Self-Guided.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention participants will receive a theory-based mHealth intervention that includes personalized nutrition and physical activity goals, psychoeducation, and evidence-based behavioral skills training delivered via a mobile web app with active content during the first 6 months, provision of digital tools to facilitate self-monitoring (a smart scale and physical activity tracker), an individual video kick-off session, text messages, and access to a closed social networking group with moderated prompts from study staff to foster peer support. Participants are encouraged to log in to web app daily to interact with self-monitoring and behavioral guidance instruction, activities, and feedback.
  Interventions: Behavioral: AYA WELL Intervention
- Self-Guided (Active Comparator): Self-guided participants will receive digital tools (a smart scale and activity tracker), an individual video kick-off session, quarterly informational newsletters, and a moderated but non-prompted (by study staff) closed social networking group to enable peer support.
  Interventions: Behavioral: Self-Guided

INTERVENTIONS:
Behavioral: AYA WELL Intervention — Behavioral weight management intervention for adolescent and young adult cancer survivors with digital tools, smartphone web app behavioral program, text messages, and expert-guided closed social networking group for peer support.
  Arms: Intervention
Behavioral: Self-Guided — Self-guided intervention with digital tools, periodic informational support, and moderated social networking group for peer support.
  Arms: Self-Guided

SUMMARY:
The AYA WELL study is a 2-arm randomized clinical trial to test the efficacy of a theory-based, mHealth weight management intervention adapted specifically for adolescent and young adult cancer survivors compared to a self-guided arm. Participants, diagnosed with cancer between ages 15-39, currently age 18-39, post-treatment at least 6 months, and who have overweight or obesity will be randomized to receive either: 1) a comprehensive mHealth weight management program (intervention) or 2) digital tools + health education + peer support (self-guided) over 12 months. Outcomes will be assessed at 3, 6, and 12 months.

DETAILED DESCRIPTION:
AYA WELL is a multi-site randomized clinical trial to test the efficacy of a 6-month theory-based, mHealth weight management intervention designed specifically for adolescent and young adult (AYA) cancer survivors, compared to a self-guided arm. The intervention is grounded in self-determination theory and designed to promote intrinsic motivation for behavior change by enhancing perceived competence, relatedness, and autonomy. The mHealth intervention includes personalized nutrition and physical activity goals, psychoeducation, evidence-based behavioral skills training, digital tools to facilitate self-monitoring (smart scale and activity tracker), tailored feedback, text messages, and access to a closed social networking group to foster peer support. The self-guided arm will receive digital tools, education, and a social networking group for peer support. The 6-month intervention will be followed by a 6-month maintenance phase (peer support only). AYA survivors (N=240, diagnosed between ages 15-39 [current age 18-39], posttreatment >6 months, body mass index [BMI] 25-50 kg/m2) will be randomized to: 1) mHealth intervention or 2) self-guided (digital tools + education + peer support only). Randomization will be stratified by BMI, sex assigned at birth, and race/ethnicity. Assessments will occur at 0 (baseline), 3 (intervention mid-point), 6 (post-intervention), and 12 months (follow-up). Percent weight change at 6 months (primary outcome) will be assessed using a remote data collection protocol via fasted video weigh-in via smart scale to facilitate enhanced reach across the US. Secondary outcomes include frailty (frailty index), objectively measured physical activity (Fitbit), dietary intake (ASA24), and quality of life (SF-36), as well as validated surveys assessing hypothesized psychosocial mediators targeted by the intervention. A subsample of participants will complete in-person visits at each clinical site (UNC and VCU) at 0, 6, and 12 months to assess changes in body composition, waist circumference, frailty, and biomarkers of aging and cardiometabolic disease. Specific aims are:

AIM 1: To test the efficacy of a theory-based, mHealth weight management intervention compared with a self-guided control arm on percent weight change among AYA cancer survivors.

AIM 2: To determine the efficacy of the intervention compared to self-guided control on secondary outcomes.

AIM 3: To examine whether changes in putative theoretical mechanisms (competence, relatedness, autonomy) mediate the effects of the intervention on weight change.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years old at the time of consent.
* Diagnosed with first invasive cancer between ages 15-39 years (self-report).
* Within 10 years of diagnosis with no evidence of progressive disease or second primary cancers (self-report).
* Completed active cancer directed therapy (cytotoxic chemotherapy, radiation therapy and/or definitive surgical intervention) at least six months prior to enrollment; may be receiving "maintenance" therapy to prevent recurrences (self-report).
* Body mass index (BMI) of 25-50 kg/m2

Exclusion Criteria:

* Type 1 diabetes or currently receiving certain medical treatments for Type 2 diabetes
* Report a history of heart attack or stroke within previous 6 months
* Health problems which preclude ability to walk for physical activity (e.g., lower limb amputation). Participants endorsing items 1-4 on the Physical Activity Readiness Questionnaire (PAR-Q) (experience of heart problems, frequent chest pains, or faintness or dizziness) will be excluded from the study.
* Lost 5% or more of body weight (and kept it off) in the last 3 months
* Lifetime history of clinical diagnosis or treatment of eating disorder (anorexia nervosa or bulimia nervosa), OR report of compensatory behaviors within the previous 3 months
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 12 months
* Untreated thyroid disease or any changes (type or dose) in thyroid medication in last 6 months
* Hospitalization for depression or other psychiatric disorder within the past 12 months.
* History of psychotic disorder or uncontrolled bipolar disorder
* Currently participating in a weight loss, nutrition, or physical activity study or program or other study that would interfere with this study
* Currently using prescription medications with known effects on appetite or weight (e.g., oral steroids, weight loss medications), with the exception of individuals on a stable dose of SSRIs for 3 months)
* Previous surgical procedure for weight loss or planned weight loss surgery in the next year
* Inability to speak and read English
* Does not reside in the United States
* Do not have mobile phone with data plan or willing to be contacted by study through text messaging
* No Internet access
* Not willing to be randomized to either intervention arm

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Weight change percent | Baseline to 6 months
  Change in weight (%) from baseline to 6 months. Weight will be objectively measured on a digital scale in the participant's home for remote participants and in the clinic for in person assessments. Percent weight change at 6 months is calculated as ((weight (kg) at 6 months - weight (kg) at baseline)/(weight (kg) at baseline))*100.

SECONDARY OUTCOMES:
Weight maintenance percent | 6 to 12 months
  Weight will be objectively measured on a digital scale in the participant's home for remote participants and in the clinic for clinic subsample. Percent weight change at 6 months is calculated as ((weight (kg) at 6 months - weight (kg) at baseline)/(weight (kg) at baseline))*100. Maintenance of weight change is measured from 6 to 12 months.
Body Mass Index (BMI) | Baseline up to 12 months
  Change in body mass index is calculated as weight in kg divided by the square of height in meters. BMI is calculated at each weight assessment and change over time is assessed.
Health-related quality of life | Baseline up to 12 months
  Change in health-related quality of life is measured using the Medical Outcomes Study 36-Item Short Form (SF-36) survey. This survey includes 36 items with eight subscales (physical functioning, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions). Responses are coded on a scale of 0 to 100, where 0 is the worst possible health and 100 is the most favorable health score. The coded responses will be summed to yield a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score. The measure is administered at baseline, 3, 6, and 12 months and change over time is assessed.
Diet quality | Baseline up to 12 months
  Diet Quality id assessed using the Healthy Eating Index (HEI) using data from the National Cancer Institute's Automated Self-Administered 24-hour Recall (ASA-24). The ASA24 measures food intake for 24 hours and calculates the HEI. Scores for the HEI range from 0 to 100. A higher score represents a better outcome. Participants complete a weekday and weekend day recall at baseline, 6, and 12 months and change over time is assessed.
Device-measured physical activity | Baseline up to 12 months
  Change in physical activity is measured as a sum of weekly minutes of light and moderate-to-vigorous physical activity at 6 and 12 months compared to baseline, assessed via wrist-worm Fitbit device. Participants are asked to wear the Fitbit device for a one week during each assessment period at baseline, 6, and 12 months. Change in weekly active minutes will be assessed over time.
Self-reported physical activity | Baseline up to 12 months
  Physical activity will be assessed using the Paffenbarger Physical Activity Questionnaire (PAQ) which assesses leisure-time activity. The PAQ provides an estimate of minutes per week of moderate-to-vigorous intensity, and calories/week of light (5 kcal/min), medium (7.5 kcal/min), and high (10 kcal/min) intensity activities. PAQ changes have been predictive of weight change. The measure is administered at baseline, 6, and 12 months and change over time is assessed.
Frailty Index | Baseline up to 12 months
  Frailty will be assessed among all participants with a Frailty Index (all participants) Five items assess self-reported fatigue (from SF-36), weight loss, morbidities, difficulty with ambulation (PROMIS Global Health), and ability to overcome resistance (from SF-36).181 The number of positive responses for these components is summed to create the FRAIL index (range 0-5). A value > 3 is considered frail, and a value of 2 is considered prefrail. Frailty is measured at baseline, 6, and 12 months and change over time is assessed.
Frailty Phenotype | Baseline up to 12 months
  Frailty will be assessed in a subset of participants assessed in person with a modified Fried frailty phenotype. The modified Fried frailty phenotype includes five clinically derived factors: 1) weakness (sitting dominant hand-grip strength using hand-held dynamometer and BMI-specific cut points); 2) slowness (timed 15-foot walk); 3) sarcopenia (relative mass of =1.5 SDs below age-, sex-, race-specific values from NHANES using bioelectrical impedance analysis; 4) exhaustion (vitality subscale of SF-36; and 5) low energy expenditure (<383 kcal/week for males, < 270 kcal/week for females from Paffenbarger Physical Activity Questionnaire). Individuals with 3 factors are classified as frail and those with 2 factors as pre-frail. Frailty is measured at baseline, 6, and 12 months and change over time is assessed.
p16 Expression | Baseline up to 12 months
  Peripheral blood will be collected from a subset of participants assessed in-person. Samples will be used to measure expression of T lymphocyte p16. At each assessment, a whole blood sample of 8mL will be drawn and collected into a 8mL ACD tube. From the ACD tube, analysis of p16 expression will be measured using a TaqMan quantitative reverse-transcription polymerase chain reaction (RTPCR) performed by Sapere Bio (Research Triangle Park, NC). The measure is collected at baseline, 6, and 12 months and change over time will be assessed.
Biomarkers of cardiovascular disease | Baseline up to 12 months
  Fasting blood samples (after an overnight fast of at least 8 hours) will be collected from a subset of participants assessed in person. At each assessment, a whole blood sample (collected in one 8.5 mL SST tube) will be collected, processed to serum, and analyzed by LabCorp for lipids (total cholesterol, HDL-C, LDL-C and triglycerides), glucose, and insulin levels. The measures are collected at baseline, 6, and 12 months and change over time will be assessed.
Blood pressure | Baseline up to 12 months
  Blood pressure will be assessed in a subset of participants assessed in person with a calibrated blood pressure monitor. Cuff size will be determined by arm circumference. After a 5-minute rest period and with both feet flat on floor, three readings will be taken, with 60 seconds between measurements. The measurement is collected at baseline, 6, and 12 months and change in systolic and diastolic blood pressure will be assessed over time.
Waist circumference | Baseline up to 12 months
  Waist circumference will be assessed in a subset of participants assessed in person, measured at the midpoint between highest point of iliac crest and lowest point of costal margin using a Gulik tape measure and following a standard protocol. Two measures of waist circumference are taken; if the difference exceeds 0.5 cm, a third measure is taken. The measurement is collected at baseline, 6, and 12 months and change over time will be assessed.
Body composition assessed by Air Displacement Plesthymography | Baseline up to 12 months
  Body composition assessed in a subset of participants with the BodPod (COSMED USA, Inc.). Participants are asked to fast for 8 hours (including caffeine) and to refrain from strenuous exercise for 8 hours prior to these body composition measures. Outcome variable of interest is change in the ratio of lean muscle mass to fat mass. The measurement is collected at baseline, 6, and 12 months and change in the ratio of lean muscle mass to fat mass is assessed over time.
Accelerometer measured physical activity | Baseline up to 12 months
  Physical activity will be assessed among the subset of participants completing in-person assessments using ActiGraph accelerometers (GT3X+, Pensacola, FL), which provides an objective assessment to corroborate self-report PA and sedentary activity data. Participants will be instructed to wear the device at all times for a full week; monitoring for at least 600 min/day for at least 5 days in the week (including at least one weekday and one weekend day) is considered adequate for analysis. Data will be aggregated into sedentary, light and MVPA using standard thresholds. Physical activity with accelerometer will be assessed at baseline, 6, and 12 months.

OTHER OUTCOMES:
Depressive Symptoms | Baseline up to 12 months
  The Center for Epidemiological Studies Depression Scale (CES-D) will be used to examine levels of depressive symptoms. The CES-D is a self-report scale designed to measure depression symptoms in the general population. The self-test measure includes 20 items that relate to depressive feelings and behaviors during the past week. Items are scored on a range of 0 (rarely or none of the time) to 3 (most or all of the time) with values ranging from 0 to 60. Higher values indicate more depressive symptoms. The measure is administered at baseline, 3, 6, and 12 months and change over time is assessed.
Perceived Stress | Baseline up to 12 months
  The 10-item Perceived Stress Scale (PSS-10) measures overall perceived stress during the past month. Items are scored on a 5-point Likert scale from 0 (Never) to 4 (Very Often) with total scores ranging from 0 to 40. Items 4, 5, 7 and 8 are reverse scored. Higher scores indicate higher levels of perceived stress. The measure is administered at baseline, 3, 6, and 12 months and change over time is assessed.
Anxiety | Baseline up to 12 months
  The Generalized Anxiety Disorder 7-item scale (GAD-7) is a self-report measure of generalized anxiety symptoms.183 Possible scores range from 0 to 21, with higher scores reflecting greater symptom severity; cut-points of 5, 10, and 15 correspond to mild, moderate, and severe levels of anxiety. The measure is administered at baseline, 3, 6, and 12 months and change over time is assessed.
Global Health | Baseline up to 12 months
  The patient-reported outcomes measurement information system (PROMIS) Global Health measure be used to measure perceptions of health. The PROMIS measure consists of 10 self-reported global health items, which assess 5 domains: physical function, pain, fatigue, emotional distress, and social health. The response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. Higher values indicate better health. The measure is administered at baseline, 3, 6, and 12 months and change over time is assessed.
Competence | Baseline up to 12 months
  Change in perceived competence from baseline to 3, 6 and 12 months as measured using the Perceived Competence for Scale. The Scale measures perceived competence for diet (4 items) and physical activity (4 items). Items are rated on a 7-point Likert scale (1 = not at all true, 7 = very true), and include items such as "I feel confident in my ability to maintain a healthy diet." Scores are summed for the items in the subscale (diet and physical activity) and the range for each subscale is 4 - 28. Greater values indicate higher levels of perceived competence for engaging in positive diet and physical activity behaviors. Scores are summed for the items in the subscale (diet and physical activity). Competence is a hypothesized mediator in this study.
Relatedness | up to 12 months
  Relatedness will be measured with 3 items adapted from the 8-item Relatedness subscale of the Basic Need Satisfaction at Work Scale. Examples include "The program demonstrates caring about me as a person" and are scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree). Responses are averaged with a range of 1 to 7. Higher scores indicate a higher level of perceived relatedness from the intervention messages. The measure will be administered at 3, 6, and 12 months and change over time will be assessed. Relatedness is a hypothesized mediator in this study.
Autonomy Support | up to 12 months
  Items are adapted from the Health Care Climate Questionnaire, which is a measure of how the participant perceives support from a healthcare provider, to measure autonomy support from the program. The scale includes 15 items rated on a scale of 1 (strongly disagree) to 7 (strongly agree) (e.g., "I feel that [the program] has provided me choices and options.") Scores are calculated by averaging the individual item scores (with item 13 reverse-scored). Higher average scores represent a higher level of perceived autonomy support. Autonomy support will be measured at 3, 6, and 12 months. Autonomy Support is a hypothesized mediator in this study.
Autonomous Motivation | Baseline up to 12 months
  Change in treatment self-regulation from baseline to 3, 6, and 12 months as measured using the Treatment Self-Regulation Questionnaire (TSRQ). The TSRQ assesses autonomous and controlled motivation for making changes in diet (15 items) and physical activity (15 items). Examples item: "Because I feel that I want to take responsibility for my own health" answered on a scale of 1 (not at all true) to 7 (very true)." Calculating the scores for the sub-scales will consist of averaging the items on that subscale. They are: Autonomous Regulation: 2, 3, 7, 10, 13, 16, 18, 19 Controlled Regulation: 1, 4, 5, 6, 8, 9, 11, 12, 14, 15, 17. Responses to the items within the subscale are averaged with the range of scores being 1 to 7. Higher values on each subscale indicate greater levels of that type of motivation. Autonomous Motivation is a hypothesized mediator in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Carmina G. Valle, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Jessica Gokee LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data sharing will be under the auspices of UNC-approved data-sharing agreements with investigators wishing to use the data. Specific requests will provide a limited dataset to prospective investigators after any data-cleaning prior to sharing. Potential investigators will submit a request to the Contact PI (Valle) that includes hypotheses, variables needed, and plans for disseminating findings.
  Final research data analyzed for publication of main trial findings as specified in our specific aims will be made available no later than acceptance of data for publication. Any publication will be embargoed per the journal's requirements or regulations and will be made publicly available no later than 12 months after the official date of publication in accordance with NIH Public Access Policy. The release of specific data may be delayed if data are part of an analysis being prepared for a separate publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning at 12 and continuing for 36 months following publication
Access Criteria: Investigator has UNC PI-approved proposal, institutional IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC